CLINICAL TRIAL: NCT04037748
Title: A Prospective, Single Dose, Randomized, Open-label, Crossover, Comparative Study to Establish Bioequivalence in Healthy Subjects Between the Puran T4® (Sanofi Aventis Farmacêutica Ltda) vs. the New Formulation of Levothyroxine (Eutirox NF® Merck) Administered Orally as 3 Tablets of 200 μg
Brief Title: Bioequivalence of Two Formulations of Levothyroxine Sodium 200 Micrograms (mcg) Under Tablet Form
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200125_0014
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-08

CONDITIONS: Healthy
Keywords: Eutirox®; Puran T4®; Levothyroxine
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Puran T4®, then Eutirox® (Experimental): Participants received single oral dose of Puran T4® 600 micrograms (mcg) (3 tablets of 200 mcg Levothyroxine sodium) in Treatment Period 1 followed by single oral dose of Eutirox® 600 mcg (3 tablets of 200 mcg Levothyroxine sodium) in Treatment Period 2 under fasting conditions. A wash-out period of 70 days was maintained between the Treatment Periods 1 and 2.
  Interventions: Drug: Puran T4®; Drug: Eutirox®
- First Eutirox®, then Puran T4® (Experimental): Participants received single oral dose of Eutirox® 600 mcg (3 tablets of 200 mcg Levothyroxine sodium) in Treatment Period 1 followed by single oral dose of Puran T4® 600 mcg (3 tablets of 200 mcg Levothyroxine sodium) in Treatment Period 2 under fasting conditions. A wash-out period of 70 days was maintained between the Treatment Periods 1 and 2.
  Interventions: Drug: Puran T4®; Drug: Eutirox®

INTERVENTIONS:
Drug: Puran T4® — Participants who received a single oral dose of Puran T4® 600 mcg tablets (3 tablets of 200 mcg Levothyroxine sodium) in either Treatment Period 1 or 2 under fasting conditions.
Drug: Eutirox® — Participants who received a single oral dose of Eutirox® 600 mcg tablets (3 tablets of 200 mcg Levothyroxine sodium) in either Treatment Period 1 or 2 under fasting conditions.

SUMMARY:
The study was to verify if the test formulation of Levothyroxine sodium presents an equivalent rate and extension of absorption to the comparator formulation when administered with the same dosage and under fasting conditions and after baseline correction concentrations.

ELIGIBILITY:
Inclusion Criteria:

* To have freely agreed and signed the consent form, after all essential elements of the protocol have been clarified, before any procedure
* Body Mass Index (BMI) of the research participants must be comprised within the range of 18.50 to 27.00
* No abnormal findings on medical history that, in the opinion of the investigator, constitutes a risk or a contraindication for the participation of the participant in the study or that could interfere with the study objectives, conduct or evaluation
* Normal vital signs: heart rate between 50 and 100 beats per minute; Systolic pressure between 80 and 129 millimeters of mercury (mmHg); diastolic pressure between 50 and 89 mmHg; temperature between 36.0 and 37.0 degrees Celsius
* Electrocardiogram (ECG) normal (abnormalities, even if clinically not relevant, are not permitted [example {e.g.}: PR, QRS, QT, QTcF] should be within normal range, no conduction abnormalities etcetera [etc.])
* All values for biochemistry and hematology tests of blood and urine within the normal range or showing no clinically relevant deviation as judged by the Investigator
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Supplementary tests results out of the values considered as normal, unless considered clinically irrelevant
* Research participants who are submitted to surgery before the beginning of the study will be carefully evaluated by the doctor regarding the enrollment in the study complying to an exclusion period ranging from 4 to 8 weeks
* Positive test for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) in pre-study tests
* Participants with a history of hypersensitivity/allergy to study drug or excipients, history or presence of asthma or any serious allergy (requiring hospitalization or prolonged systemic treatment), any food allergy or intolerance which in the opinion of the Investigator represents a safety risk (e.g., iodine allergy, etc.)
* Has participated in any experimental trial or has taken any experimental drug within 6 months previous to this study (RDC [resolution of the collegiate board] Resolution 34, dated June 3, 2008)
* Participants that prior to the dosing takes any other medication and had not passed at least seven half-lives of elimination of the drug, in this case, be considered by the Principal Investigator the non-inclusion of the participant in the study. Participants taking medications known to affect thyroid hormone metabolism, e.g., oral contraceptives, hormonal implants, parenteral hormones, anabolic steroids, androgens, etc., or the bioavailability of levothyroxine like proton pump Inhibitors
* Has a history of alcohol abuse or has ingested alcohol 24 hours previous to the hospitalization period
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Instituto de Ciências Farmacêuticas de Estudos e Pesquisas, Aparecida de Goiânia, Brazil

IPD SHARING:
Plan to Share IPD: No
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany, will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.merckgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200125_0014
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | First Puran T4®, Then Eutirox® | First Eutirox®, Then Puran T4®
Started | 36 | 36
Completed | 28 | 30
Not Completed | 8 | 6
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 4 | 5
Period: Treatment Period 2
Arm/Group | First Puran T4®, Then Eutirox® | First Eutirox®, Then Puran T4®
Started | 28 | 30
Completed | 26 | 29
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First Puran T4®, Then Eutirox® | First Eutirox®, Then Puran T4® | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.0 (8.7) | 35.9 (9.3) | 35.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 18 | 18 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Baseline Corrected Maximum Observed Plasma Concentration (Cmax[Adj]) of Levothyroxine Sodium
Description: Cmax was obtained from plasma concentration time curve. Maximum plasmatic concentration observed adjusted by basal level correction was reported.
Time Frame: Pre-dose, 24, 36, 48 and 72 hours post-dose
Population: Pharmacokinetic (PK) analysis set included all participants who completed both periods and had valid PK parameters in both.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Puran T4® | Eutirox®
Number analyzed (Participants) | 55 | 55
Nanogram per milliliter (ng/mL) | 67.258 (19.654) | 60.552 (13.61)
Statistical Analysis 1: Comparison: Puran T4® vs Eutirox®; Test type: Equivalence — Bio-equivalence Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Geometric least squares (LS) mean ratio = 90.8, 90% CI 2-sided [86.3 to 95.6]

2. Primary Outcome: Baseline Corrected Area Under The Plasma Concentration-time Curve From Time Zero to 72 Hours (AUC0-72 [Adj]) of Levothyroxine Sodium
Description: The AUC 0-72 was defined as the area under the plasma concentration versus time curve from time zero (pre-dose) to 72 hours post-dose. Area under the plasma curve from time 0 hours to time 72 hours adjusted by basal levels correction was reported.
Time Frame: Pre-dose, 24, 36, 48 and 72 hours post-dose
Population: PK analysis set included all participants who completed both periods and had valid PK parameters in both.
Measure: Mean (Standard Deviation); unit: Hour* ng/mL
Arm/Group | Puran T4® | Eutirox®
Number analyzed (Participants) | 55 | 55
Hour* ng/mL | 2682.371 (795.263) | 2516.055 (716.575)
Statistical Analysis 1: Comparison: Puran T4® vs Eutirox®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 93.7, 90% CI 2-sided [88.2 to 99.5]

3. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Levothyroxine Sodium
Description: Tmax was obtained from plasma concentration time curve.
Time Frame: Pre-dose, 24, 36, 48 and 72 hours post-dose
Population: PK analysis set included all participants who completed both periods and had valid PK parameters in both.
Measure: Median (Full Range); unit: Hours
Arm/Group | Puran T4® | Eutirox®
Number analyzed (Participants) | 55 | 55
Hours | 3.50 [1.00 to 6.00] | 4.00 [1.50 to 8.00]

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 72 Hours (AUC 0-72) of Levothyroxine Sodium
Description: The AUC 0-72 was defined as the area under the plasma concentration versus time curve from time zero (pre-dose) to 72 hours post-dose.
Time Frame: Pre-dose, 24, 36, 48 and 72 hours post-dose
Population: PK analysis set included all participants who completed both periods and had valid PK parameters in both.
Measure: Mean (Standard Deviation); unit: Hour* ng/mL
Arm/Group | Puran T4® | Eutirox®
Number analyzed (Participants) | 55 | 55
Hour* ng/mL | 7204.615 (1337.674) | 7004.507 (1154.596)
Statistical Analysis 1: Comparison: Puran T4® vs Eutirox®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 97.3, 90% CI 2-sided [94.7 to 100.0]

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Levothyroxine Sodium
Description: Cmax was obtained from plasma concentration time curve.
Time Frame: Pre-dose, 24, 36, 48 and 72 hours post-dose
Population: PK analysis set included all participants who completed both periods and had valid PK parameters in both.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Puran T4® | Eutirox®
Number analyzed (Participants) | 55 | 55
ng/mL | 130.069 (25.464) | 122.895 (18.957)
Statistical Analysis 1: Comparison: Puran T4® vs Eutirox®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 94.82, 90% CI 2-sided [92.0 to 97.8]

ADVERSE EVENTS:
Time Frame: Up to 79 Days; Participants were assessed for adverse events for the entire study.
Description: Safety analysis set included all randomized participants who received one dose of study drug.
Groups:
- Puran T4: Participants who received a single oral dose of Puran T4® 600 mcg tablets (3 tablets of 200 mcg Levothyroxine sodium) in either Treatment Period 1 or 2 under fasting conditions.
Arm/Group | Puran T4 | Eutirox®
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 2/72 | 5/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Puran T4 (N=72) | Eutirox® (N=72)
Vomiting (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 3
Lipothymia (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT04037748/Prot_SAP_000.pdf